CLINICAL TRIAL: NCT07178314
Title: Evaluating the Feasibility and Efficacy of At-Home Transcutaneous Tibial Nerve Stimulation (TTNS) for Overactive Bladder in Rural Women
Brief Title: At-Home Transcutaneous Tibial Nerve Stimulation for Overactive Bladder in Rural Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Principal Investigator, Sara Cichowski, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028373
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Overactive Bladder
Keywords: Transcutaneous Tibial Nerve Stimulation (TTNS); Rural Healthcare
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: All study participants will receive the intervention.
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rural Women Treated with Transcutaneous Tibial Nerve Stimulation (Experimental): Participants will undergo a self-implemented at-home Transcutaneous Tibial Nerve Stimulation (TTNS) treatment protocol for management of treatment naive overactive bladder (OAB) among rural dwelling women.
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation (TTNS)

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation (TTNS) — Participants will perform self-implemented at-home transcutaneous tibial nerve stimulation using a transcutaneous electrical nerve stimulation (TENS) unit. Participants will be instructed to use the TENS unit to deliver stimulation to the tibial nerve on one ankle for a 30-minute session, three times per week for 12 weeks upon receipt of the device. Intensity will be based on the participant's tolerance, just above the perception threshold but not painful.
  Other Names: TTNS; TENS Unit

SUMMARY:
This study contains a mixed-methods design consisting of a single-arm, interventional study and prospective patient interviews evaluating a novel self-implemented at-home Transcutaneous Tibial Nerve Stimulation (TTNS) treatment protocol for management of treatment naïve overactive bladder (OAB) among rural-dwelling women. This study will be conducted in 3 rural Oregon communities where Oregon Health & Science University satellite campuses are located.

DETAILED DESCRIPTION:
A total of 38 participants who meet the inclusion criteria will be recruited from clinical sites in three rural Oregon counties: 1) Klamath County, 2) Jefferson County, and 3) Coos County. Potential subjects with overactive bladder (OAB) who are being seen at healthcare clinics including primary care, obstetrics and gynecology, and pelvic floor physical therapy will be informed of this research study. Interested participants will be referred to the study coordinator via a flyer. Participants will be screened by phone and if deemed eligible and elect to participate, they will be consented over the phone/web platform. The participant has the option to sign a paper consent should they not have access to the internet. This will be mailed to them with prepaid postage for return of the signed consent. If a person does not elect to participate, the study team will offer the person information about behavioral modifications for treatment of overactive bladder and/or a referral to a local pelvic floor physical therapist. All communication and patient facing information will be offered in English or Spanish, utilizing Oregon Health & Science University's (OHSU's) interpreter services for translation from English as described above.

Our intervention focuses on self-implemented at-home transcutaneous tibial nerve stimulation (TTNS) using a transcutaneous electrical nerve stimulation (TENS) unit. The TENS device is a nonsignificant risk device. A TENS unit with preset settings, labeled device, reusable electrodes, a battery, and detailed instructions will be mailed to the participant's designated address. All participants will receive a set of written instructions in the mail with details on skin preparation, application of the two electrodes to their ankle, connection of the electrodes to the TENS unit, standardized stimulation parameters, and adjustment of intensity to perception threshold. The written instructions will contain pictures and graphics that guide correct placement of the electrodes and use of the TENS unit settings. All participants will also be provided with a link to a short video demonstrating the application and use of the TENS unit. The script for this video is submitted with this IRB application.

Our protocol will instruct participants to use the TENS unit to deliver stimulation to the tibial nerve on one ankle for a 30-minute session, three times per week for 12 weeks starting treatment upon receipt of the device. The standardized stimulation parameters include pulse frequency of 10 Hz and pulse width of 200 ms, as used in previous studies. The intensity level is based on the participant's tolerance, ideally just above the perception threshold but not painful. Participants will be contacted by telephone at 2-3 week intervals to check on compliance with the protocol and address any issues. They will be given the study team's contact information to call sooner if questions or issues arise. Participants will also be provided with an electronic or printed 12 week calendar to keep track of completed sessions.

All participants recruited into the interventional study will also be approached and consented for possible involvement in individual interviews at their initial enrollment. Following completion of the intervention, the PI and co-investigator will use purposive sampling to identify 10-20 key informants for one-on-one video and/or audio recorded interviews with a member of the research group. Informants in the study sample are selected by investigators considering several parameters including demographic features, baseline and post-intervention scores on questionnaires from the primary and secondary outcomes previously mentioned, and compliance rate. Key informant interviews will provide insights on participant's unique experiences with self-managed TTNS at home, allowing for determination of patient perceived facilitators and barriers to this intervention. These key topics and themes can be used to inform future practices regarding self-implemented TTNS among rural dwelling patients.

A list of pre-determined, open-ended questions will be asked to each participant addressing different themes. The script and questions for the interview portion will be submitted alongside this proposal. Interviews will be recorded and transcribed verbatim using software licensed through the OHSU library (Dedoose). The software will be utilized to identify key themes emerging from the interview process. Data collection will cease once thematic saturation has been achieved, determined by the PI and co-investigator.

ELIGIBILITY:
Inclusion Criteria:

* Rural residence (as defined by the Federal Office of Rural Health policy confirmed with the "Am I rural?" tool)
* Clinical diagnosis of overactive bladder (OAB) with urinary frequency >= 8 times per day
* Able to complete questionnaires, urination diaries, and interview in English or Spanish
* Have reliable access to a telephone or email for communication
* Ambulatory and able to use the toilet independently

Exclusion Criteria:

* Unable to consent
* Pregnancy or planning to become pregnant during the study period
* Previous treatment for OAB including medication, intravesical botox, and/or neuromodulation use
* Presence of pacemaker or implantable defibrillator
* Indwelling metal in both ankles
* Presence of leg ulcers, open wounds, or skin conditions affecting lower legs
* Absence of sensation in the lower legs
* Active urinary tract infection
* Predominantly stress urinary incontinence
* Active malignancy
* Neurogenic bladder
* Subjective complaint of pelvic organ prolapse outside of vaginal introitus
* Subjective symptoms of incomplete bladder emptying
* Epilepsy
* Peripheral artery disease affecting both legs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder questionnaire short form (OAB-q SF) Health-related Quality of life | Evaluated upon enrollment and following 12 weeks of intervention
  A 13-item survey assessing health-related quality of life. Assessed on a scale from 1 to 100 with a higher score representing a better quality of life.
Overactive Bladder questionnaire short form (OAB-q SF) symptom bother | Evaluated upon enrollment and following 12 weeks of intervention
  A 13-item survey assessing symptom bother related to overactive bladder. Assessed on a scale from 1 to 100 with a higher score representing more bother, which is a worse outcome.
24-hour voiding frequency | 3-day voiding diary completed upon enrollment and following 12 weeks of intervention
  Mean 24-hour voiding frequency based on a 3-day voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cichowski, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States